CLINICAL TRIAL: NCT00474617
Title: A Multicenter, Parallel Group, Comparative, Phase IIIa Trial to Compare the Efficacy, Safety, and Pharmacokinetics of Org 25969 in Elderly Subjects With Adult Subjects
Brief Title: Comparison of the Efficacy, Safety, and Pharmacokinetics of Sugammadex (MK-8616; Org 25969) in Elderly Participants With Adult Participants (MK-8616-029)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05950; 19.4.305 (Other: Organon Study Number); P05950 (Other: Schering-Plough Study Number); MK-8616-029 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Results first posted 2019-03-25 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Participants 18 to 64 years old (Experimental): Participants to receive an intravenous (IV) single bolus dose of 0.6 mg.kg-1 rocuronium. If further neuromuscular block was required after endotracheal intubation, maintenance dose(s) of 0.15 mg.kg-1 rocuronium were to be administered. After the intubation dose or the last maintenance dose of rocuronium, participants were to be reversed at reappearance of second twitch (T2) with an intravenous single bolus dose of 2.0 mg.kg-1 of sugammadex.
  Interventions: Drug: Sugammadex; Drug: Rocurium
- Participants 65 to 74 years old (Experimental): Participants to receive an IV single bolus dose of 0.6 mg.kg-1 rocuronium. If further neuromuscular block was required after endotracheal intubation, maintenance dose(s) of 0.15 mg.kg-1 rocuronium were to be administered. After the intubation dose or the last maintenance dose of rocuronium, participants were to be reversed at reappearance of T2 with an intravenous single bolus dose of 2.0 mg.kg-1 of sugammadex.
  Interventions: Drug: Sugammadex; Drug: Rocurium
- Participants 75 years and older (Experimental): Participants to receive an IV single bolus dose of 0.6 mg.kg-1 rocuronium. If further neuromuscular block was required after endotracheal intubation, maintenance dose(s) of 0.15 mg.kg-1 rocuronium were to be administered. After the intubation dose or the last maintenance dose of rocuronium, participants were to be reversed at reappearance of T2 with an intravenous single bolus dose of 2.0 mg.kg-1 of sugammadex.
  Interventions: Drug: Sugammadex; Drug: Rocurium

INTERVENTIONS:
Drug: Sugammadex
  Other Names: Org 25969; MK-8616
Drug: Rocurium — intravenous (IV) single bolus dose of 0.6 mg.kg-1

SUMMARY:
The purpose of the study is to compare the effectiveness, safety and pharmacokinetics of sugammadex in participants 65 and over with participants under 65. There is no hypothesis defined for the study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class 1 to 3
* 18 years of age or older
* Scheduled for elective surgical procedure under general anesthesia requiring neuromuscular block with the use of rocuronium
* Scheduled for surgery in supine position
* Given written informed consent

Exclusion Criteria:

* Participants in whom a difficult intubation is expected due to anatomical malformations
* Participants known or suspected to have neuromuscular disorders impairing neuromuscular blockade and/or significant renal dysfunction
* Participants known or suspected to have a (family) history of malignant hyperthermia
* Participants known or suspected to have an allergy to narcotics, muscle relaxants or other medications used during surgery
* Participants receiving medication known to interfere with neuromuscular blocking agents such as anticonvulsants, antibiotics and magnesium
* Female participants who are pregnant or breast-feeding
* Females participants of childbearing potential not using an acceptable method of birth control [condom or diaphragm with spermicide, vasectomized partner (> 6 months), intrauterine device (IUD), abstinence]
* Participants who had already participated in a Org 25969 trial including Protocol 19.4.305
* Participants who had participated in another clinical trial, not pre-approved by Organon, within 30 days of entering into Protocol 19.4.305

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2005-12-29 (Actual); Primary Completion 2006-10-20 (Actual); Study Completion 2006-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] McDonagh DL, Benedict PE, Kovac AL, Drover DR, Brister NW, Morte JB, Monk TG. Efficacy, safety, and pharmacokinetics of sugammadex for the reversal of rocuronium-induced neuromuscular blockade in elderly patients. Anesthesiology. 2011 Feb;114(2):318-29. doi: 10.1097/ALN.0b013e3182065c36. PMID 21239968
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants 18 to 64 Years Old: Participants to receive an IV single bolus dose of 0.6 mg.kg-1 rocuronium. If further neuromuscular block was required after endotracheal intubation, maintenance dose(s) of 0.15 mg.kg-1 rocuronium were to be administered. After the intubation dose or the last maintenance dose of rocuronium, participants were to be reversed at reappearance of second twitch (T2) with an intravenous single bolus dose of 2.0 mg.kg-1 of sugammadex.
Period: Overall Study
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Started | 56 | 64 | 42
Treated | 48 | 62 | 40
Completed | 48 | 61 | 40
Not Completed | 8 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for all participants that received study drug.
Groups:
- Participants 18 to 64 Years Old: Participants to receive an intravenous IV single bolus dose of 0.6 mg.kg-1 rocuronium. If further neuromuscular block was required after endotracheal intubation, maintenance dose(s) of 0.15 mg.kg-1 rocuronium were to be administered. After the intubation dose or the last maintenance dose of rocuronium, participants were to be reversed at reappearance of T2 with an intravenous single bolus dose of 2.0 mg.kg-1 of sugammadex.
- Total: Total of all reporting groups
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older | Total
Number analyzed (Participants) | 48 | 62 | 40 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (11.32) | 69.2 (2.53) | 80.1 (4.08) | 64.5 (15.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 24 | 80
  Male | 19 | 35 | 16 | 70

OUTCOME MEASURES:

1. Primary Outcome: Mean Time From Start of Administration of Sugammadex to Recovery of the T4/T1 Ratio to 0.9
Description: Neuromuscular function was monitored by applying repetitive train-of-four (TOF) electrical stimulations with the TOF-Watch® SX to the ulnar nerve of one forearm every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 are the magnitudes (heights) of the first and fourth twitches respectively after TOF nerve stimulation, where stimulation was continued until the T4/T1 ratio reached 0.9. A higher T4/T1 ratio indicates a lower degree of neuromuscular blockade, with a value of 1.0 representing full recovery.
Time Frame: up to 10 minutes from start of sugammadex
Population: All participants that received study drug and had at least 1 post-baseline efficacy measurement. Missing data were imputed.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Participants 18 to 64 Years Old; Participants 65 to 74 Years Old; Participants 75 Years and Older: Participants to receive an IV single bolus dose of 0.6 mg.kg-1 rocuronium. If further neuromuscular block was required after endotracheal intubation, maintenance dose(s) of 0.15 mg.kg-1 rocuronium were to be administered. After the intubation dose or the last maintenance dose of rocuronium, participants were to be reversed at reappearance of T2 with an intravenous single bolus dose of 2.0 mg.kg-1 of sugammadex.
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 48 | 62 | 40
Minutes | 2.53 (1.35) | 2.92 (1.63) | 3.93 (1.67)

2. Secondary Outcome: Mean Time From Start of Administration of Sugammadex to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular function was monitored by applying repetitive train-of-four (TOF) electrical stimulations with the TOF-Watch® SX to the ulnar nerve of one forearm every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 are the magnitudes (heights) of the first and fourth twitches respectively after TOF nerve stimulation, where stimulation was continued until the T4/T1 ratio reached 0.7. A higher T4/T1 ratio indicates a lower degree of neuromuscular blockade, with a value of 1.0 representing full recovery.
Time Frame: up to 10 minutes from start of sugammadex
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 48 | 62 | 40
Minutes | 1.77 (0.78) | 2.10 (1.47) | 2.68 (1.17)

3. Secondary Outcome: Mean Time From Start of Administration of to Recovery of the T4/T1 Ratio to 0.8
Description: Neuromuscular function was monitored by applying repetitive train-of-four (TOF) electrical stimulations with the TOF-Watch® SX to the ulnar nerve of one forearm every 15 seconds & assessing twitch response at the adductor pollicis muscle. T1 and T4 are the magnitudes (heights) of the first and fourth twitches respectively after TOF nerve stimulation, where stimulation was continued until the T4/T1 ratio reached 0.8. A higher T4/T1 ratio indicates a lower degree of neuromuscular blockade, with a value of 1.0 representing full recovery.
Time Frame: up to 10 minutes from start of sugammadex
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 48 | 62 | 40
Minutes | 2.05 (0.98) | 2.38 (1.55) | 3.10 (1.35)

4. Secondary Outcome: Participants Level of Consciousness Prior to Transfer to the Recovery Room After Extubation
Description: Participants level of consciousness was assessed post-extubation and prior to transfer to recovery room. The levels were reported as: awake and oriented; arousable with minimal stimulation; responsive only to tactile stimulation. The number of participants in each of the 3 categories was summarized.
Time Frame: Prior to Transfer to the Recovery Room After Extubation (up to 24 hours)
Population: All participants that received study drug, had at least 1 post-baseline efficacy measurement and had data available for endpoint.
Measure: Number; unit: Participants
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 47 | 61 | 40
Participants
  Awake and oriented | 24 | 38 | 21
  Arousable with minimal stimulation | 21 | 22 | 17
  Responsive only to tactile stimulation | 2 | 1 | 2

5. Secondary Outcome: Participants Level of Consciousness Prior to Discharge From Recovery Room
Description: Participants level of consciousness was assessed prior to discharge from the recovery room. The levels were reported as: awake and oriented; arousable with minimal stimulation; responsive only to tactile stimulation. The number of participants in each of the 3 categories was summarized.
Time Frame: Prior to Discharge from Recovery Room (up to 24 hours)
Population: All participants that received study drug and had at least 1 post-baseline efficacy measurement and had data available for endpoint
Measure: Number; unit: Participants
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 46 | 58 | 38
Participants
  Awake and oriented | 43 | 56 | 36
  Arousable with minimal stimulation | 3 | 2 | 2
  Responsive only to tactile stimulation | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With General Muscle Weakness Prior to Transfer to the Recovery Room After Extubation
Description: The number of participants experiencing general muscle weakness was assessed by the investigator as a measure of recovery from neuromuscular blockade post-extubation and prior to transfer to recovery room. A standardized examination form was used to determine the presence or absence of muscle weakness in various muscle groups and the overall assessments were reported as "yes" or "no" to general muscle weakness. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Prior to Transfer to the Recovery Room After Extubation (up to 24 hours)
Population: All participants that received study drug, had at least 1 post-baseline efficacy measurement and were determined to be cooperative.
Measure: Number; unit: Participants
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 45 | 60 | 34
Participants | 0 | 3 | 1

7. Secondary Outcome: Number of Participants With General Muscle Weakness Prior to Discharge From Recovery Room
Description: The number of participants experiencing general muscle weakness was assessed by the investigator as a measure of recovery from neuromuscular blockade prior to discharge from the recovery room. A standardized examination form was used to determine the presence or absence of muscle weakness in various muscle groups and the overall assessments were reported as "yes" or "no" to general muscle weakness. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Prior to Discharge from Recovery Room (up to 24 hours)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 46 | 58 | 38
Participants | 0 | 0 | 1

8. Secondary Outcome: Number of Participants Who Can Perform a 5 Second Head Lift Prior to Transfer to the Recovery Room After Extubation
Description: Participants were asked to lift their head off the table while in a supine position post-extubation and prior to transfer to recovery room. The number of participants who could perform the 5 second head lift was summarized. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Prior to Transfer to the Recovery Room After Extubation (up to 24 hours)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 45 | 60 | 34
Participants | 40 | 57 | 31

9. Secondary Outcome: Number of Participants Who Can Perform a 5 Second Head Lift Prior to Discharge From Recovery Room
Description: Participants were asked to lift their head off the table while in a supine position just prior to discharge from the recovery room. The number of participants who could perform the 5 second head lift was summarized. Participants who were not cooperative with the examination were not included in the assessment.
Time Frame: Prior to Discharge from Recovery Room (up to 24 hours)
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
Number analyzed (Participants) | 46 | 58 | 38
Participants | 46 | 58 | 38

ADVERSE EVENTS:
Time Frame: up to 7 days after administration of the study drug
Description: Population included all participants that received study drug.
Arm/Group | Participants 18 to 64 Years Old | Participants 65 to 74 Years Old | Participants 75 Years and Older
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/62 | 0/40
Serious Adverse Events (participants affected / at risk) | 4/48 | 8/62 | 3/40
Other Adverse Events (participants affected / at risk) | 48/48 | 62/62 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants 18 to 64 Years Old (N=48) | Participants 65 to 74 Years Old (N=62) | Participants 75 Years and Older (N=40)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1)
Abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter related complication (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants 18 to 64 Years Old (N=48) | Participants 65 to 74 Years Old (N=62) | Participants 75 Years and Older (N=40)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 7 (7) | 5 (5)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 7 (7) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (14) | 16 (16) | 15 (16)
Vomiting (Gastrointestinal disorders) | 7 (7) | 9 (9) | 5 (5)
Chills (General disorders) | 1 (1) | 3 (3) | 4 (4)
Oedema peripheral (General disorders) | 1 (1) | 4 (4) | 3 (4)
Pyrexia (General disorders) | 5 (6) | 11 (12) | 6 (6)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Incision site complication (Injury, poisoning and procedural complications) | 4 (5) | 3 (3) | 0 (0)
Post procedural nausea (Injury, poisoning and procedural complications) | 9 (9) | 6 (6) | 3 (3)
Procedural hypertension (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 44 (49) | 57 (63) | 36 (41)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 8 (8) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 5 (5)
Headache (Nervous system disorders) | 8 (8) | 3 (3) | 7 (7)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in the protocol will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.